CLINICAL TRIAL: NCT02991352
Title: Stereotactic MRI Based Image Guidance for the Treatment of Vascular Malformations - a Pilot Study
Acronym: SIGVaM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3193; 2016-00827 (Other: Kantonale Ethikkommission Bern (KEK))
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Vascular Malformations
Keywords: Vascular Malformations; Image Guidance
MeSH Terms: conditions — Vascular Malformations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Image guided needle placement into vascular malformations based on MRI
  Interventions: Device: Image guided needle placement

INTERVENTIONS:
Device: Image guided needle placement — Stereotactic MRI based image guidance to aid in the placement of percutaneous needles into vascular malformations using a CE marked navigation system (CAS-One IR, CAScination AG)

SUMMARY:
Treatment of vascular malformations requires the placement of a needle within anatomically non well defined, pathological vessels, which may be as small as 1 mm, with the current state of the art relying exclusively on two dimensional fluoroscopy images for guidance. The investigators hypothesize that the combination of stereotactic image guidance with existing targeting methods will result in faster and more reproducible needle placements.

DETAILED DESCRIPTION:
This prospective study aims to investigate the feasibility of the utilization of stereotactic image guidance technology for the needle based percutaneous treatment of peripheral vascular malformations. The specific device to be utilized is the CAS-One IR system, CE marked for use with needle based procedures in combination with medical image data including MRI data, as required by this study.

Utilizing feedback from the stereotactic image guidance system, the interventionalist will attempt to place the needle within the malformation. The position and orientation of the needle relative to the anatomy will be displayed on 2D slices from the MRI, as well as relative to a 3D volume rendering of the patient anatomy constructed from MRI data. The position of the needle relative to the desired position within the malformation will be evaluated utilizing fluoroscopy.

If necessary the position of the needle will be adjusted, this adjustment can be performed utilizing navigated feedback or standard fluoroscopy feedback at the discretion of the physician. The final position of the needle will be confirmed on intra-operative DSA imaging and the sclerosant will be applied according to standard clinical protocols.

This single-centre pilot study will involve a total of 10 patients suffering from peripheral vascular malformations. Only non-emergency adult patients will be considered for inclusion in this trial. Inclusion will be at the discretion of the treating physician and patient. As the study is designed as a pilot trial, no comparator is considered and no blinding performed. The trial will be performed over a period of nine months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with venous or mixed venous-lymphatic malformation
* Patients which are regular scheduled for a percutaneous treatment of a vascular malformation
* Informed Consent as documented by signature

Exclusion Criteria:

* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2017-11-29 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Time to reach the target | During the intervention (duration approx. 90 minutes on average)
  Time from start of targeting to alcohol embolization in minutes

SECONDARY OUTCOMES:
Radiation time | During the intervention (duration approx. 90 minutes on average)
  Measured by the C-arm imaging device in seconds
Radiation dose | During the intervention (duration approx. 90 minutes on average)
  Measured by the C-arm imaging device in μGym²
Contrast agent volume | During the intervention (duration approx. 90 minutes on average)
  Measured by the nurses in milliliter
Number of attempts | During the intervention (duration approx. 90 minutes on average)
  Defined as number of skin punctures, counted by the investigator
Reason to change to standard approach | During the intervention (duration approx. 90 minutes on average)
  Asked by the investigator
System Usability Score (SUS) | Directly after the intervention (60 minutes afterwards at the latest)
  Filled out by the interventionalist

CONTACTS AND LOCATIONS:
Overall Officials: Iris Baumgartner, MD, Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (3):
- Switzerland (3):
  - ARTORG Center for Biomedical Engineering, Bern
  - Universitätsinstitut für Diagnostische, Interventionelle und Pädiatrische Radiologie, Bern
  - Universitätsklinik für Angiologie, Bern

IPD SHARING:
Plan to Share IPD: No